CLINICAL TRIAL: NCT01995708
Title: A Phase I Trial of Vaccination With CT7, MAGE-A3, and WT1 mRNA-electroporated Autologous Langerhans-type Dendritic Cells as Consolidation for Multiple Myeloma Patients Undergoing Autologous Stem Cell Transplantation
Brief Title: CT7, MAGE-A3, and WT1 mRNA-electroporated Autologous Langerhans-type Dendritic Cells as Consolidation for Multiple Myeloma Patients Undergoing Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-009
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: CT7; MAGE-A3; WT1 mRNA-electroporated Autologous Langerhans; vaccine; Autologous Stem Cell Transplantation; 13-009
MeSH Terms: conditions — Multiple Myeloma | interventions — MAGEC1 protein, human; MAGEA3 protein, human; Standard of Care

ARMS (2):
- Arm 1 Vaccine (Experimental): This is a prospective, two-arm phase I randomized trial. Patients will be accrued only from and treated at MSKCCand The Rockefeller University/Center for Clinical & Translational Science . The study will assess autologous LCs presenting CT7, MAGE-A3, and WT1 after electroporation with CT7, MAGE-A3, and WT1 mRNA. Twenty patients will accrue to the study and ten will receive vaccines at 9x10^6 LCs per dose (i.e., combination of 3x10^6 CT7 mRNA-electroporated LCs + 3x10^6 MAGE-A3 mRNA-electroporated LCs + 3x10^6 WT1 mRNA-electroporated LCs) and another ten who will not receive any LC vaccines but will otherwise undergo identical cytoreduction, ASCT, and standard supportive care. At approximately 3 months after ASCT and as deemed clinically appropriate, patients will start lenalidomide maintenance therapy, which is now standard to delay disease progression.
  Interventions: Biological: CT7, MAGE-A3, and WT1 mRNA-electroporated Langerhans cells ( LCs)
- Arm 2 control (Active Comparator): Patients receive standard of care treatment after autologous stem cell transplant
  Interventions: Other: Standard of care

INTERVENTIONS:
Biological: CT7, MAGE-A3, and WT1 mRNA-electroporated Langerhans cells ( LCs) — Patients receive CT7/MAGE-A3/WT1 mRNA-electroporated autologous Langerhans-type dendritic cells ID on days 12, 30, and 90 after autologous stem cell transplant. Patients on the vaccine arm of the study will receive a total of 3 vaccinations, comprising a primary immunization on day +12 after ASCT followed by two boosters at days +30 and +90. Vaccines will be dosed at 9x10^6 LCs per vaccine x 3.
  Arms: Arm 1 Vaccine
Other: Standard of care — No vaccines
  Arms: Arm 2 control

SUMMARY:
The purpose of this study is to see if the investigator can help the immune system to work against myeloma.

This study will see if a vaccine made with altered dendritic cells will make T cells work against tumor cells. The stem cells collected for the transplant will also be used to grow dendritic cells in the lab. The dendritic cells will carry the antigens. These cells then will be injected under the skin. The investigators will do lab studies before and after the vaccination to find out if the vaccine is working.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma, ISS stages I-III, within 12 months of starting therapy.
* Completion of induction therapy with Very Good Partial Response (VGPR), or better, by International Myeloma Working Group (IMWG) criteria.
* Deemed eligible for ASCT by standard institutional criteria.
* Age ≥18 years.
* Documentation of CT7, MAGE-A3, or WT1 expression in the bone marrow and/or bone marrow aspirate.

Exclusion Criteria:

* Prior autologous or allogeneic SCT.
* Previous immunization against CT7, MAGE-A3, other cancer-testis antigens, or WT1.
* Known immunodeficiency, HIV positivity, hepatitis B, or hepatitis C.
* History of autoimmune disease (e.g., rheumatoid arthritis, SLE), other than vitiligo, diabetes, or treated thyroiditis, which are allowed.
* History of severe allergic reactions to vaccines or unknown allergens.
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first immunization.
* Lenalidomide-related toxicities before ASCT necessitating its discontinuation as part of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chung, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Chung DJ, Sharma S, Rangesa M, DeWolf S, Elhanati Y, Perica K, Young JW. Langerhans dendritic cell vaccine bearing mRNA-encoded tumor antigens induces antimyeloma immunity after autotransplant. Blood Adv. 2022 Mar 8;6(5):1547-1558. doi: 10.1182/bloodadvances.2021005941. PMID 35100339
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 Vaccine | Arm 2 Control
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Vaccine | Arm 2 Control | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Median (Full Range); unit: years] | 58 [46 to 68] | 62 [51 to 68] | 59 [46 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 10 | 14 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 10 | 14 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for Vaccine Safety
Description: Participants will be evaluated for the safety of the vaccine, monitored and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0 for toxicity and adverse event reporting to the Food and Drug Administration. Dose limiting toxicity (DLT) is defined as grade 3 or higher toxicity. The only toxicities captured outside of the SAEs reported will be all grade 1-5 toxicites deemed definitely, probably, or possibly related to the vaccine portion of the study.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Vaccine | Arm 2 Control
Number analyzed (Participants) | 13 | 15
Participants | 13 | 15

2. Secondary Outcome: Median Progression Free Survival
Description: Median profression free survival.
Time Frame: Up to 7 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 Vaccine | Arm 2 Control
Number analyzed (Participants) | 13 | 15
months | 31 [3 to 63] | 54 [12 to 85]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm 1 Vaccine | Arm 2 Control
All-Cause Mortality (participants affected / at risk) | 12/13 | 8/15
Serious Adverse Events (participants affected / at risk) | 3/13 | 2/15
Other Adverse Events (participants affected / at risk) | 13/13 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Vaccine (N=13) | Arm 2 Control (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Vaccine (N=13) | Arm 2 Control (N=15)
Anemia (Blood and lymphatic system disorders) | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 5
Lymphocyte count decreased (Investigations) | 10 | 11
Neutrophil count decreased (Investigations) | 7 | 11
Platelet count decreased (Investigations) | 10 | 10
White blood cell decreased (Investigations) | 10 | 11
Lung infection (Infections and infestations) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT01995708/Prot_SAP_000.pdf